CLINICAL TRIAL: NCT00981864
Title: A Feasibility Study to Evaluate Intensity Modulated Radiation Therapy (IMRT) for Concomitant Boost Breast Radiotherapy (CBRT)
Brief Title: Concurrent Boost Radiotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 07-0594-C
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: radiation therapy in breast cancer; concurrent radiation; Breast cancer patients
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Concurrent Boost RT (Experimental)
  Interventions: Radiation: Concurrent Boost RT

INTERVENTIONS:
Radiation: Concurrent Boost RT — Patient will receive radiation to the tumour bed concurrently with whole breast radiation instead of receiving this treatment sequentially, that is, whole breast RT first then followed by RT directly to the tumour bed.

SUMMARY:
The primary aim of this study is to evaluate the feasibility of delivering 42.5 Gy to the breast with a concomitant 10 Gy boost to the tumour bed in 16 fractions for a total duration of 3.5 weeks using intensity modulated radiotherapy (IMRT). The primary end-point is the proportion of patients treated without major treatment deviation.

DETAILED DESCRIPTION:
Rather than a sequential boost, we propose delivering a concomitant boost using intensity modulated radiotherapy (IMRT). IMRT is a sophisticated technique deliberately using multiple non-uniform beams, resulting in complex, conformal dose distributions. This technique offers several advantages. A concomitant IMRT boost potentially offers improved dose distributions by allowing more conformal doses around the boost volume and increased sparing of the remaining breast and adjacent organs at risk. Several studies have shown better target dose homogeneity resulting in less toxicity with adjuvant breast IMRT . One study found a significant reduction in the rates of moist desquamation with IMRT compared to wedged tangential fields (31% vs. 48%, P=0.0014).

Longer treatment duration increases the inconvenience and decreases patient compliance. Furthermore, this places extra financial and emotional hardship on the patient and her family, particularly if they must travel long distances between home and the treatment centre. Studies have found 10-30% of patients do not receive adjuvant radiotherapy after lumpectomy,placing these patients at higher risk for local recurrence and death from disease. Radiobiologically, a boost increases the risk of late normal tissue effects. In the EORTC study, they found significantly higher but limited rates of severe fibrosis at 10 years of 4.4% vs. 1.6% (p<0.0001) with the boost. No age effect was noted on the incidence of fibrosis. One study compared a shorter hypofractionated schedule of 42.5 Gy/16 fractions over 3.5 weeks with the standard schedule of 50 Gy/25 fractions over 5 weeks and observed comparable 5 year local recurrence rates and cosmetic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient with a new histological diagnosis of invasive carcinoma OR ductal carcinoma-in-situ (DCIS) of the breast and no evidence of metastatic disease.
2. Any of the following indications for boost radiotherapy to tumour bed:

   1. Age ≤ 60 years
   2. Positive or close resection margins (≤ 2 mm)
   3. Lymphovascular space invasion
   4. Extensive intraductal component (DCIS >25% of tumour volume)
3. Three or fewer axillary nodes involved as determined either by:

   1. Sentinel node biopsy OR
   2. Axillary node dissection OR
   3. Clinical exam for patients with DCIS only or age greater than 70 years of age.
4. Informed consent.

Exclusion Criteria:

1. Age < 18 years.
2. Seroma or surgical cavity on CT estimated to be > 30% of the breast volume.
3. More than one primary tumour in different quadrants of the same breast.
4. Previous irradiation to the ipsilateral breast that would preclude whole breast irradiation.
5. Presence of an ipsilateral breast implant or pacemaker.
6. Serious non-malignant disease (e.g. cardiovascular, pulmonary, systemic lupus erythematosus (SLE), scleroderma) which would preclude definitive radiation treatment.
7. For patients not treated with adjuvant chemotherapy: unable to commence radiation therapy within 12 weeks of the last surgical procedure on the breast.
8. For patients treated with adjuvant chemotherapy: unable to commence within 8 weeks of the last dose of chemotherapy.
9. Previous or concomitant malignancies except for patients with nonmelanoma skin cancer, contralateral non-invasive breast cancer or carcinoma in situ of any other site. In addition, patients with invasive cancers treated more than 5 years previously and without evidence of recurrence will be eligible.
10. Currently pregnant or lactating.
11. Psychiatric or addictive disorders which would preclude obtaining informed consent or adherence to protocol.
12. Geographic inaccessibility for follow-up.
13. Regional lymphatic irradiation planned.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of delivering 42.5 Gy to the breast with a concomitant 10 Gy boost to the tumour bed in 16 fractions without major treatment deviation. | 2 years

SECONDARY OUTCOMES:
To evaluate acute and late morbidity related to treatment | 2 years
To identify factors and parameters associated with increased risk of treatment morbidity | 2 years
To evaluate local control rates | 2 years
To develop treatment protocol outlining appropriate guidelines for planning and delivery | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fei-Fei Liu, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada